CLINICAL TRIAL: NCT02784353
Title: Clinical Outcomes of Preoperative and Postoperative Rehabilitation in the Patients With HBP(Hepatobiliary and Pancreatic) Malignancy
Brief Title: Clinical Outcomes of Preoperative and Postoperative Rehabilitation in the Patients With HBP Malignancy
Acronym: PReHeBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae Wook Hwang, Assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PReHeBP; 2015-665 (Other Grant/Funding Number: Asan Medical Center)
Record Dates: First submitted 2016-05-06; First posted 2016-05-27 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Hepatic Neoplasms; Biliary Tract Neoplasms; Pancreatic Neoplasms
Keywords: Rehabilitation; Quality of life; Surgery; Hepatic neoplasms; Biliary tract neoplasms; Pancreatic neoplasms
MeSH Terms: conditions — Liver Neoplasms; Biliary Tract Neoplasms; Pancreatic Neoplasms | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: 2 arm, parallel, randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The result of allocation in control and intervention group would be blinded to primary and secondary outcomes assessor.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Active Comparator): No intervention; conventional perioperative management without perioperative rehabilitation program
  Interventions: Behavioral: Conventional
- Intervention - PReHeBP (Experimental): conventional perioperative management with preoperative and postoperative rehabilitation program
  Interventions: Behavioral: Perioperative rehabilitation program

INTERVENTIONS:
Behavioral: Perioperative rehabilitation program — Perioperative rehabilitation program
  * preoperative rehabilitation : 2 weeks prior to operation
  * postoperative rehabilitation : 3 months after operation
  Other Names: PReHeBP
  Arms: Intervention - PReHeBP
Behavioral: Conventional — conventional perioperative management without rehabilitation program
  Other Names: No intervention
  Arms: Conventional

SUMMARY:
Clinical Outcomes of Preoperative and Postoperative Rehabilitation in the Patients With HBP Malignancy.

DETAILED DESCRIPTION:
The most important outcome in the management of HBP malignancies is survival. Since the application of ERAS (enhanced recovery after surgery), the improvement of QOL(quality of life) has been known as one of important factor for the management of HBP malignancies as well as survival, and the improvement of QOL, itself, affect the survival.

There are several reports that perioperative rehabilitation affect positively for the outcome of surgery and QOL in surgical patients. However, in the HBP field, there are rarely studied for this concept.

This study aim to investigate that the application of rehabilitation program for the surgery of HBP malignancies affect on short-term outcome and lead the improvement of QOL.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old or <80 years old
* ECOG 0-2
* resectable HBP malignancies or premalignant lesions which should be required GI resection and anastomosis
* open surgery
* no distant metastasis
* no functional disturbance in bone marrow; WBC at least 3,000/mm3 or absolute neutrophil count at least 1,500/mm3, Platelet count at least 125,000/mm3
* no functional disturbance in liver; AST less than 5 times upper limit of normal
* no function disturbance in kidney; Creatinine no greater than 1.5 times upper limit of normal
* informed consent

Exclusion Criteria:

* distant metastasis (+) or recurred HBP tumor
* active or uncontrolled infection
* alcohol or other drug addiction
* already enrolled patient in other study which affect this study
* pregnant or the possibility of pregnancy (+)
* uncontrolled cardiopulmonary disease
* moderate to severe comorbidity which affect on the quality of life and nutritional status (liver cirrhosis, end stage renal disease, heart failure, etc.)
* previous history of major gastrointestinal surgery (gastrectomy, colectomy, etc.)
* previous history of neurological or musculoskeletal diseases which is impossible to allow investigator's order

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of general complication | till postoperative 3 months
  Incidence rate and severity of general complications except operation-specific complication, according to Clavien-Dindo classification

SECONDARY OUTCOMES:
The incidence of operation-specific complication | till postoperative 3 months
  Incidence rate and severity of operation-specific complication, according to Clavien-Dindo classification
The incidende of Mortality | till postoperative 3 months
  Rate of in-hospital mortality and 90 days mortality
Rate of re-admission | till postoperative 3 months
  the rate of re-admission, till postoperative 3 months
The changes in Quality of life | Comparison between at the time of discharge and postoperative 3months
  changes in quality of life (EORTC QLQ-C30), at the time of discharge and 3 months after surgery
Compliance of Aerobic exercise, strength exercise and respiratory excursion (Changes in the parameters of rehabilitation) | Initial(2 weeks before surgery), preoperative (within 2days prior to surgery) and 3 months after surgery
  Compliance of Aerobic exercise, strength exercise and respiratory excursion based on exercise diary
Measurement on 6 minutes walk test (m/minute) (Changes in the parameters of rehabilitation) | Initial(2 weeks before surgery), preoperative (within 2days prior to surgery) and 3 months after surgery
  Measure the 6 minutes walk test (m/minute)
Grasping power(dynamometer, kg)(Changes in the parameters of rehabilitation) | Initial(2 weeks before surgery), preoperative (within 2days prior to surgery) and 3 months after surgery
  Grasping power measurement using dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: DAE WOOK HWANG, M.D., Principal Investigator — Asan Medical Center, University of Ulsan College of Medicine, SEOUL, KOREA
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831
- [Result] Ford-Smith CD, Wyman JF, Elswick RK Jr, Fernandez T. Reliability of stationary dynamometer muscle strength testing in community-dwelling older adults. Arch Phys Med Rehabil. 2001 Aug;82(8):1128-32. doi: 10.1053/apmr.2001.24291. PMID 11494194
- [Result] Johansson K, Tibe K, Weibull A, Newton RC. Low intensity resistance exercise for breast cancer patients with arm lymphedema with or without compression sleeve. Lymphology. 2005 Dec;38(4):167-80. PMID 16515225
- [Result] Otsuji H, Yokoyama Y, Ebata T, Igami T, Sugawara G, Mizuno T, Nagino M. Preoperative sarcopenia negatively impacts postoperative outcomes following major hepatectomy with extrahepatic bile duct resection. World J Surg. 2015 Jun;39(6):1494-500. doi: 10.1007/s00268-015-2988-6. PMID 25651963
- [Result] Schwartz AL. Fatigue mediates the effects of exercise on quality of life. Qual Life Res. 1999 Sep;8(6):529-38. doi: 10.1023/a:1008978611274. PMID 10548868
- [Result] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Result] Yeo TP, Burrell SA, Sauter PK, Kennedy EP, Lavu H, Leiby BE, Yeo CJ. A progressive postresection walking program significantly improves fatigue and health-related quality of life in pancreas and periampullary cancer patients. J Am Coll Surg. 2012 Apr;214(4):463-75; discussion 475-7. doi: 10.1016/j.jamcollsurg.2011.12.017. Epub 2012 Feb 7. PMID 22321518
- [Result] Yun YH, Park YS, Lee ES, Bang SM, Heo DS, Park SY, You CH, West K. Validation of the Korean version of the EORTC QLQ-C30. Qual Life Res. 2004 May;13(4):863-8. doi: 10.1023/B:QURE.0000021692.81214.70. PMID 15129896
- [Result] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Result] Bobbio A, Chetta A, Ampollini L, Primomo GL, Internullo E, Carbognani P, Rusca M, Olivieri D. Preoperative pulmonary rehabilitation in patients undergoing lung resection for non-small cell lung cancer. Eur J Cardiothorac Surg. 2008 Jan;33(1):95-8. doi: 10.1016/j.ejcts.2007.10.003. Epub 2007 Nov 19. PMID 18006327
- [Result] Wittes J, Brittain E. The role of internal pilot studies in increasing the efficiency of clinical trials. Stat Med. 1990 Jan-Feb;9(1-2):65-71; discussion 71-2. doi: 10.1002/sim.4780090113. PMID 2345839